CLINICAL TRIAL: NCT00353769
Title: A Single-blinded Comparative Study on Hair Apposition Technique Performed Between Nurses and Doctors in Emergency Department.(HAT2 Study)
Brief Title: Comparison Study on Hair Apposition Technique Performed Between Nurses and Doctors in Emergency Department.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: DCR/P15/2003
Record Dates: First submitted 2006-07-17; First posted 2006-07-19 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Scalp Laceration
Keywords: scalp laceration; tissue adhesive; wound care; cost effectiveness

INTERVENTIONS:
Procedure: Hair Apposition Technique

SUMMARY:
The purpose of this study is to compare the effectiveness, complications and benefits of Hair Apposition Technique(HAT)performed by nurses or doctors.

DETAILED DESCRIPTION:
Hair Apposition Technique (HAT) is a relatively new technique for treating certain scalp lacerations. It has been shown to be equally acceptable as compared to the standard toilet and suture. This procedure has been the technique of choice for suitable scalp lacerations in Department of Emergency Medicine, Singapore General Hospital (DEM, SGH) and Emergency Medicine Department, National University Hospital (EMD, NUH).

Currently HAT is being performed by doctors in the respective hospitals. Nurses, on the other hand, are routinely using tissue adhesives for minor wound closure. However, nurses in Kandang Kerbau Women and Children Hospital (KKWCH) have been routinely using HAT for 1 year now. Studies had been also been done by nurses in treating of minor wounds using various tissue adhesives as well as hair knotting technique.The trend of nurses handling minor wounds with tissue adhesives, hair knotting technique as well as HAT suggested the possibility of nurses performing HAT to a degree as competent as a doctor.

This study aims to compare the effectiveness, complications and benefits HAT performed between nurses and doctors in the Emergency Department.

ELIGIBILITY:
Inclusion Criteria:

* All age group
* Linear lacerations of scalp
* Lacerations less than 10cm in length
* Hair at least 3cm in length

Exclusion Criteria:

* Severely contaminated wounds
* Actively bleeding wounds
* Patients with unstable vital signs or altered mental state

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 360
Dates: Start 2002-11; Study Completion 2005-02

PRIMARY OUTCOMES:
Presence of any complications, namely infection, scarring, bleeding, wound breakdown and allergy
Satisfactory wound healing

SECONDARY OUTCOMES:
Duration of procedure
Pain perception

CONTACTS AND LOCATIONS:
Overall Officials: Ong EH Marcus, M.D, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore